CLINICAL TRIAL: NCT02965677
Title: Evaluation of the Safety and Efficacy of the Paclitaxel Releasing Peripheral Balloon Dilatation Catheter （LEGFLOW）in Treatment of Stenosis or Occlusion in Femoral-popliteal Arteries：A Prospective, Multicenter, Randomized, Controlled Clinical Study
Brief Title: A Study of The Femoral Popliteal Artery Treated With LEGFLOW OTW
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ZhuHai Cardionovum Medical Device Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LEGFLOW-2015-01
Record Dates: First submitted 2016-11-07; First posted 2016-11-17 (Estimated); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Peripheral Arterial Disease
Keywords: drug eluting balloon; Femoral Popliteal Artery
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LEGFLOW OTW group (Experimental): in this group subject will be treated by Paclitaxel Releasing Peripheral Balloon Dilatation Catheter (LEGFLOW) and followed up
  Interventions: Device: Paclitaxel Releasing Peripheral Balloon Dilatation Catheter
- Admiral Xtreme (Active Comparator): in this group subject will be treated by Peripheral Balloon Dilatation Catheter (Admiral Xtreme) and followed up
  Interventions: Device: Peripheral Balloon Dilatation Catheter

INTERVENTIONS:
Device: Paclitaxel Releasing Peripheral Balloon Dilatation Catheter — in this group the subject will be treated by Paclitaxel Eluting Balloon Dilatation Catheter
  Other Names: LEGFLOW OTW
  Arms: LEGFLOW OTW group
Device: Peripheral Balloon Dilatation Catheter — in this group the subject will be treated by Paclitaxel Eluting Balloon Dilatation Catheter
  Other Names: Admiral Xtreme
  Arms: Admiral Xtreme

SUMMARY:
To evaluate the safety and efficacy of the Paclitaxel Releasing Peripheral Balloon Dilatation Catheter (LEGFLOW) compared with the standard balloon (Admiral Xtreme) for the treatment of stenosis or occlusions in femoral popliteal artery.

DETAILED DESCRIPTION:
To evaluate the safety and efficacy of the Paclitaxel Releasing Peripheral Balloon Dilatation Catheter (LEGFLOW) compared with the standard balloon (Admiral Xtreme) for the treatment of stenosis or occlusions in femoral popliteal artery.

This is a prospective, multicenter, prior desiged, randomize and controlled study, planned to enrol 172 subjects. all these subjects will be allocated 1:1 to the LEGFLOW OTW group n=86 and Admiral Xtreme group n=86. and accept the treatment of LEGFLOW and Admiral Xtreme balloon. and followed up at day 0-30, month 6, 12 by DUS and clinical examination. all the endpoint data will be assessed by DUS core-lab, CEC, then be statisticed.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and ≤ 85 years.
2. De novo or restenotic lesions in the femoral popliteal artery due to atherosclerosis, which located in the superficial femoral artery and/or proximal popliteal artery (arterial segment starting at least 1cm beyond the common femoral artery bifurcation to the distal P1 segment of the popliteal artery at the level of the proximal edge of the patella). And the patients are suitable for endovascular therapy with LEGFLOW OTW or Admiral Xtreme.
3. Rutherford class 2 to 5.
4. Target lesion length ≤ 200mm.
5. Target lesion stenosis ≥ 70% or total occlusion, and it can be passed with common manipulation.
6. Reference vessel diameter ≥ 4mm and ≤ 8mm by visual estimate.
7. Target lesion consists of a single of de novo or restenotic lesion, or a adjacent lesion or a combination lesion or multiple lesion which meets the following criteria:

   * adjacent lesion: (1) lesion space ≤ 30mm; (2) total lesion length (include lesion space) ≤ 200mm; (3) can be treated as a single lesion.
   * Combination lesion: combination lesion is defined as not a chronic total occlusion (CTO), but may include a part of total occlusion (100% stenosis). The total lesion length ≤ 200mm.
   * Multiple lesion: (1) lesion space > 30mm; (2) total lesion length (include lesion space) ≤ 200mm; (3) can be treated as multiple lesions.
8. Angiographic evidence of adequate distal run-off to the foot (at least one native calf vessel is patent, defined as < 50% diameter stenosis), whether or not this outfolw was re-established by previous intervention.
9. If subject has ipsilateral/contralateral iliac disease that requires treatment during the procedure, the iliac lesions must meet all the following criteria:

   * Iliac lesion or occlusion is ≤ 100mm in length;
   * must be treated before the target lesion (superficial femoral artery/proximal popliteal artery).
   * must be successfully treated before target lesion treatment; success is defined as: (1) residual stenosis < 30%; (2) free of dissection which can limit blood flow; (3) no occurrence of thrombus, embolization, or other SAE.
10. Life expectancy more than one year.
11. Understands the study objective and is willing to participate and provide the informed consent form, and is willing to comply with specified follow-up evaluations at the specified time points.

Exclusion Criteria:

1. Women of childbearing age with negative pregnancy test before procedure, and breastfeeding women.
2. Stroke or STEMI within 30 days prior to the procedure.
3. Either local or systemic thrombolytic therapy within 6 weeks prior to the procedure.
4. Any major surgical operation (operation class ≥ 3) or interventional therapy within 30 days prior to the procedure.
5. Any major selective surgical operation (operation class ≥ 3) or interventional therapy within 30 days prior to the procedure.
6. Restenotic lesions after DCB or bypass surgery.
7. Target limb has been previously treated with bypass surgery.
8. Guidewire must be passed through from the distal part of limb.
9. Known allergies or sensitivities to contrast agent, paclitaxel, anti-platelet, anticoagulants or thrombolytic drugs.
10. Known allergies or sensitivities to heparin, including those patients who have had a previous incidence of heparin-induced thrombocytopenia (HIT) type II.
11. Aneurysm located at the target vessel.
12. Acute or sub-acute thrombosis in the target vessel.
13. Angiographic evidence of severe calcification (defined as dense circumferential calcification that makes the target lesion non-dilatable and/or calcificatin that is present on both sides of the vessel wall and that extends more than 5 cntinuous centimeters in length within the target lesion prior to contrast injection or digital subtraction angiography).
14. The bilateral lower limb must be treated in one procedure.
15. Uncorrected bleeding disorder.
16. Renal insufficiency (serum creatinine >2.5mg/dL or renal dialysis).
17. Stenosis or occlusions due to non-atherosclerosis, such as thrombotic occlusive vasculitis or vasculitis.
18. Septicemia or bacteremia.
19. Patients with severe disease (such as severe chronic obstructive pulmonary disease, malignant tumor, dementia, etc.) or patient's physical condition may affect the compliance with this study.
20. Pre-dilation resulted in a major (≥ Grade D) flow-limiting dissection or residual stenosis > 70%.
21. Major distal amputation (above the transmetatarsal) in the study limb or non-study limb.
22. Patients who have participated in another investigational drug or device trial that has not completed the primary endpoint.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2016-12; Primary Completion 2020-12 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
clinically driven target lesion revascularization (CD-TLR) | 12 month post procedure

SECONDARY OUTCOMES:
Procedural Success | at 0-30 days
  Procedural Success defines as the blood supply of the target lesion regained after treatment, residual stenosis less than 50% and without flow-limiting dissection (≥type D) occurred.
Device Success | at 0-30 days
  Device Success defines as the device successfully delivered to the target location, inflated, deflated and withdrawn from the treated balloon inflation tube.
Clinical Success | at 0-30 days
  Clinical Success defines as operation success, and without any postoperative complication before discharge (death, lesions limb amputation, target lesion thrombosis or TVR)
Change in Rutherford classification measured | at 0-30 days, 6 months and 12 months post procedure
Change in ABI measure | at 0-30 days, 6 months and 12 months post procedure
Walking capacity assessment by Walking Impairment Questionnaire (WIQ) | at 0-30 days, 6 months and 12 months post procedure
Walking distance assessment by Six Minute Walk Test (6MWT) | 0-30 days, 6 months and 12 months post procedure compared with baseline
Quality of life assessment by EQ5D | at 0-30 days, 6 months and 12 months post procedure compared with baseline
Target lesion revascularization (TLR) | 0-30 days, 6 months and 12 months post procedure
Target vessel revascularization (TVR) | at 0-30 days, 6 months and 12 months post procedure
Thrombus at the target lesion site | 0-30 days, 6 months and 12 months post procedure
Target limb amputation rates | at 0-30 days, 6 months and 12 months post procedure
Major Adverse Event (MAE) rate which including all cause death, CD-TLR and major target limb amputation. | at 0-30 days, 6 months and 12 months post procedure
Clinical-driven target vessel revascularization (CD-TVR) rates | at 0-30 days, 6 months and 12 months post procedure
Clinical-driven target lesion revascularization (CD-TLR) rates | at 0-30 days, 6 months and 12 months post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Guo Wei, professor, Principal Investigator — Chinese PLA Genral Hospital
Locations (13):
- China (13):
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Hainan General Hospital, Haikou, Hainan
  - The First hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Beijing Anzhen Hospital, Capital Medical University, Beijing
  - Beijing Chao-yang Hospital, Capital Medical University, Beijing
  - Beijing Hospital, Beijing
  - Beijing Shijitan Hospital, Capital Medical University, Beijing
  - Fuwai Hospital, Chinese Accadamy of Medical Sciences, Beijing
  - Longhua Hospital Shanghai University of Tranditional Chinese Medicine, Shanghai
  - Shanghai Ninth people's Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Tianjin Medical University General Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: Undecided